CLINICAL TRIAL: NCT04107688
Title: Taste Perception, Salivary Proteins & the Oral Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Beverly J Tepper, Ph.D., Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13309M
Record Dates: First submitted 2019-04-25; First posted 2019-09-27 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Saliva Altered; Taste, Altered
Keywords: Oral Microbiome
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROP non-taster subjects (Experimental): This arm will comprise of PROP non-taster subjects. Subjects will use a cranberry-derived oral rinse twice a day for 11 days following a 3-day control-rinse period.
  Interventions: Other: Control; Other: CPE
- PROP super-taster subjects (Experimental): This arm will comprise of PROP super-taster subjects. Subjects will use a cranberry-derived oral rinse twice a day for 11 days following a 3-day control-rinse period.
  Interventions: Other: Control; Other: CPE

INTERVENTIONS:
Other: Control — Subjects will use plain water as an oral rinse twice a day for 3 days.
Other: CPE — Subjects will use a cranberry-derived oral rinse twice a day for 11 days.

SUMMARY:
Genetic differences in taste are believed to play an important role in food selection, especially for strong-tasting foods and beverages. The overall goal of this project is to better understand how genes that control food preferences differ among people and whether saliva composition and oral health are related to these differences.

This study examines the effects of a daily cranberry extract oral rinse on salivary protein responses and the oral microbiome (as a proxy measure of oral health). The study will be conducted in healthy adults who are presumably at high-risk (non-tasters of PROP; homozygous recessive for tas2R38 gene) or low-risk (super-taster of PROP; homozygous dominant for tas2R38 gene) of oral disease.

The specific aims are to determine if the use of cranberry polyphenol extract rinse will:

1. alter the oral microbial profile
2. induce changes in the salivary protein response
3. be associated with changes in taste and flavor perception

Participants will be screened for good overall and oral health (see inclusion/exclusion criteria below). Each subject's period of participation will be 2 weeks. Days 1-3 of the study is a run-in period. Subjects rinse with spring water 2-times/day (after brushing their teeth in the morning and evening). During days 4-14, subjects will rinse in a similar manner with a solution of cranberry-derived polyphenol extract (CPE) in spring water. Saliva will be collected from subjects in a brief session (10 min) on Days 3 and Day 14. Saliva samples will be analyzed for salivary proteins and microbial profile analysis. The purpose of this analysis is to measure the relative ratios of beneficial vs. disease-causing microbes in the mouth using 16S RNA sequencing. On each of the testing days, subjects will also evaluate food samples for standard taste and flavor attributes.

ELIGIBILITY:
Inclusion Criteria:

* PROP insensitive individuals (PROP non-tasters; homozygous recessive for tas2R38 gene)
* PROP high-sensitive individuals (PROP super-tasters; homozygous dominant for tas2R38 gene)
* Overall healthy; good oral health and hygiene routine
* Current on a routine checkup by a oral/dental health professional
* Recently underwent dental/cleaning by a oral/dental health professional
* No ongoing oral health problems
* Agree to use intervention material as prescribed
* Agree to refrain from using any other oral rinse material during the term of the study

Exclusion Criteria:

* PROP medium-taster individuals (heterozygous for tas2R38 gene)
* Taste or smell dysfunction
* Pregnant or nursing
* Oral piercings
* Smoking
* Use of medications other than birth control

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Taste and Flavor Intensity Ratings | 3 days after control intervention; 11 days after experimental intervention
  Taste and Flavor intensity ratings of cranberry juice samples will be collected 3 days after control intervention and then at the end of the experimental intervention. An end-anchored (None, Very Strong) 15 cm line scale will be used with taste and key flavor attributes.
Levels of Salivary Proteins | 3 days after control intervention; 11 days after experimental intervention
  Saliva will be collected 3 days after control intervention and then at the end of the experimental intervention. Samples will be analyzed via LCMS to establish proteomic composition before and after the intervention. Specifically, area of the ion current peaks (XIC peaks) generated will be used as a relative quantity of the salivary protein levels. The XIC peaks are proportional to the concentration of salivary proteins under constant conditions and will be used to understand the effect of the intervention on salivary protein levels.
Composition of Oral Microbiome | 3 days after control intervention; 11 days after experimental intervention
  Salivary samples will be collected 3 days after control intervention and then at the end of the experimental intervention. Samples will be analyzed for microbial composition via 16S rRNA sequencing and data used to understand changes in microbial diversity before and after the intervention. Specifically operational taxonomic units will be identified and classified at the genera level.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, Department of Food Science, New Brunswick, New Jersey, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT04107688/ICF_000.pdf